CLINICAL TRIAL: NCT01363622
Title: Zekai Tahir Burak Maternity Teaching Hospital
Brief Title: Vaspin Levels Compared With Serum Insulin and Blood Glucose Levels in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity and Teaching Hospital, Ahmet Akcay
Other Study IDs: ZTB061
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-03

CONDITIONS: Insulin Sensitivity
Keywords: Vaspin; LGA; SGA; Insulin; Blood glucose
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- SGA: SGA (small for gestational age)
- LGA: LGA (large for gestational age)
- AGA: AGA (appropriate-for-gestational-age)

SUMMARY:
The aim of this study was to investigate circulating concentrations of vaspin in fetal and neonatal samples from SGA, AGA and LGA with the respective insulin concentrations. Serum vaspin concentrations were determined by enzyme immunoassay in 22 SGA and 30 LGA and 30 AGA singleton full-term fetuses and neonates on cord blood and postnatal day 5.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy infant

Exclusion Criteria:

* sepsis
* congenital anomaly
* sick infant

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: SGA infant LGA infant AGA infant
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)